CLINICAL TRIAL: NCT04946669
Title: An Exploratory Study on the Efficacy and Safety of Abatacept in the Treatment of Refractory Dermatomyositis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Wenfeng Tan, Chief Physician, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABA-DM
Record Dates: First submitted 2021-05-17; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Dermatomyositis; Abatacept
Keywords: Refractory Dermatomyositis; Abatacept; Efficacy; Safety
MeSH Terms: conditions — Dermatomyositis | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Refractory Dermatomyositis (Experimental): Patients who have been receiving glucocorticoids in combination with at least one immunosuppressive therapy for at least 3 months and who have failed therapy or are intolerant to therapy
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Abatacept is a CTLA-4 fusion protein that inhibits T cell activation by competitively binding to CD80/CD86 and blocking the second signal. To date, Abatacept has been approved by the FDA for the treatment of three types of rheumatoid immune diseases (refractory rheumatoid arthritis, juvenile idiopathic arthritis, and active psoriatic arthritis). The international consensus of experts recommends abacepil as a second-line regimen for the treatment of refractory dermatomyositis based on the evidence of case reports. However, to date, there is no relevant report or clinical study registration information of Abatacept in the treatment of dermatomyositis.

SUMMARY:
Dermatomyositis is a heterogeneous disease characterized by involvement of the proximal muscles of the extremities. Some patients have treatment failure or intolerance to the above treatment regimens, which is called refractory dermatomyositis. Abatacept has been approved by the FDA for the treatment of three types of rheumatoid immune diseases, and the international consensus of experts recommends abacepil as a second-line regimen for the treatment of refractory dermatomyositis based on the evidence of case reports.

DETAILED DESCRIPTION:
Dermatomyositis is a heterogeneous disease characterized by involvement of the proximal muscles of the extremities. Some patients have skin, lung and other systems involved. The clinical manifestations of dermatomyositis are varied and vary from person to person, so the treatment should follow the principle of individualization. At present, glucocorticoid combined with immunosuppressants (including methotrexate, azathioprine, cyclosporine, tacrolimus, mycophoranate, cyclophosphamide, etc.) is the first choice for the treatment of dermatomyositis. Some patients have treatment failure or intolerance to the above treatment regimens, which is called refractory dermatomyositis. There has not been a large-scale study to explore the treatment regimens. Abatacept is a CTLA-4 fusion protein that inhibits T cell activation by competitively binding to CD80/CD86 and blocking the second signal. To date, Abatacept has been approved by the FDA for the treatment of three types of rheumatoid immune diseases (refractory rheumatoid arthritis, juvenile idiopathic arthritis, and active psoriatic arthritis). The international consensus of experts recommends abacepil as a second-line regimen for the treatment of refractory dermatomyositis based on the evidence of case reports. However, to date, there is no relevant report or clinical study registration information of Abatacept in the treatment of dermatomyositis. The purpose of this study was to prospectively observe the efficacy and safety of Abatacept in the treatment of refractory dermatomyositis through a controlled before and after study.

ELIGIBILITY:
Inclusion Criteria:

1. Dermatomyositis confirmed in accordance with Bohan-Peter criteria for inflammatory myopathy, or clinically free myopathic dermatomyositis according to the revised Sontheimer criteria, aged 18 years or older, regardless of gender.
2. Patients with refractory dermatomyositis, specifically defined as those who have received glucocorticoid combined with at least one immunosuppressive therapy for at least 3 months and have failed treatment or intolerance to treatment.Treatment failure was defined as improvement of 3 core parameters in the core assessment measures of iMACS <20%, or more than 2 parameters deterioration >25%.Treatment intolerance is defined as a patient experiencing side effects that require discontinuation of the drug or an underlying condition that prevents further use of the drug.Before enrollment, the dosage of glucocorticoids was <1mg/kg/day, prior use of at least one immunosuppressant (including methotrexate, azathioprine, cyclosporine, tacrolimus, mycophenolic ester and cyclophosphamide, etc.) at a stable dose >3 months.
3. If the patient has previously used biological agents, etc., the washout period shall be completed.
4. Patients or their guardians fully understand the content of this study, are willing to participate in the study, and sign the informed consent.

Exclusion Criteria:

1. Other rheumatoid immune diseases: including but not limited to rheumatoid arthritis, systemic lupus erythematosus, systemic sclerosis, Sjogren's syndrome, primary biliary cirrhosis, etc.
2. combined with other myopathy causing myopathy and myasthenia;These include neurological diseases (such as muscular dystrophy, myasthia gravis, amyotrophic lateral sclerosis, Guillain-Barre syndrome, etc.), tumors, drug effects (such as statins, etc.), infections, genetic diseases, endocrine diseases, electrolyte disorders, rhabdomyolysis, etc.
3. Patients with severe heart, liver, kidney and other important organs and blood and endocrine system lesions:Including but not limited to decompensated cardiac insufficiency, refractory hypertension and abnormal ecg, cereal third transaminase or aspertate aminotransferase more than 2 times higher than normal reference value online, renal tubular acidosis, renal interstitial lesions, renal insufficiency, serious leucopenia, severe anemia, severe thrombocytopenia and other serious diseases, such as tumor, etc.).
4. Active infection, glucocorticoid and immunosuppressive therapy may aggravate infection;Hepatitis B virus surface antigen and hepatitis C antibody were positive.Active TB patients who have been treated for active TB within the previous 3 years, or who have been screened for latent TB, and who are positive for PPD combined with T-SPOT, or positive for sputum bacteria.
5. Pregnant and lactating women, women of reproductive age who cannot guarantee contraception.
6. Patients with allergic constitution, who have been allergic to various drugs in the past.
7. Mental disorders, or other patients unable to cooperate with treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
IMACS score improved | 12 weeks after treat with Abatacept
  Improvement of 3 core parameters of disease activity in the core assessment index of IMACS over 20 percent with no more than 2 parameters deteriorating over 25 percent.
  And parameters of IMACS include Physician Global Assessment, Patient Global Assessment, Muscle strength assessment with MMT-8, Sports Ability Assessment Questionnaire, laboratory evaluation including creatine kinase, aldolase, lactic dehydrogenase and so on, Evaluation of myositis disease activity using MDAAT and appraisal of life quality.

SECONDARY OUTCOMES:
Dose of glucocorticoids used | 12 weeks after treat with Abatacept
  Dose of glucocorticoids used

OTHER OUTCOMES:
Occurrence of adverse events | 12 weeks after treat with Abatacept
  Occurrence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No